CLINICAL TRIAL: NCT01874938
Title: A Non-Randomized, Open-Label, Single-Arm, Phase 2 Study of LY2875358 in Patients With MET Diagnostic Positive, Advanced Gastric Cancer
Brief Title: A Study of LY2875358 in Participants With MET Positive, Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15007; I4C-JE-JTBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-22; First posted 2013-06-11 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — emibetuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2875358 (Experimental): LY2875358 will be administered intravenously (IV) at 2000 milligram (mg) bi-weekly in 28 day Cycle.
  Interventions: Biological: LY2875358

INTERVENTIONS:
Biological: LY2875358 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of LY2875358 in participants with MET diagnostic positive (+), advanced gastric or gastroesophageal junction (GEJ) cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of a histopathologically or cytologically confirmed local and/or advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma which is unresectable
* Have received 2 regimens of prior chemotherapies for gastric or GEJ adenocarcinoma
* Have the presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Have consent to provide a tissue sample for pre-screening
* Determined to be MET diagnostic positive based upon testing of a tumor sample obtained at any time before enrollment
* Have discontinued all previous treatments for cancer, including chemotherapy and radiotherapy, for at least 3 weeks before enrollment and have recovered from the acute effects of therapy
* Have adequate organ function
* Male participants: must agree to use a reliable method of birth control and to not donate sperm during the study and for at least 4 months following last dose of study drug or country requirements, whichever is longer
* Female participants: are women of child-bearing potential who test negative for pregnancy ≤14 days before enrollment based on a serum pregnancy test and agree to use a reliable method of birth control during the study and for 4 months following the last dose of the study drug and must also not be breastfeeding
* Have a performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have an estimated life expectancy, in the judgment of the investigator, of at least 12 weeks

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 21 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study or any other study investigating LY2875358
* Have an active fungal, bacterial, and/or known viral infection
* Have a history of New York Heart Association class ≥3, unstable angina, myocardial infarction (MI) in 6 months prior to study drug administration
* Have symptomatic central nervous system (CNS) malignancy or metastasis
* Have previous or concurrent malignancies
* Have received a liver transplant, or have liver cirrhosis with a Child-Pugh Stage of B or C
* Have corrected QT interval (QTc) of >470 millisecond (msec) on screening electrocardiogram (ECG)
* Have received previous treatment with any hepatocyte growth factor (HGF)/MET targeting therapeutics
* Have a history of radiation therapy involving more than 25% of the bone marrow. Previous radiation therapy is allowed but should have been limited and must not have included whole pelvis radiation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) Rate | 8 Weeks

SECONDARY OUTCOMES:
Proportion of Participants who Exhibit Confirmed Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR]) | Baseline to Confirmed CR or PR (Estimated up to 4 Months)
Proportion of Participants who Exhibit Stable Disease (SD) or Confirmed CR or PR (Disease Control Rate [DCR]) | Baseline to Measured Progressive Disease or Death from Any Cause (Estimated up to 4 Months)
Duration of Response | Date of CR or PR to Date of Measured Recurrent or Progressive Disease or Death from Any Cause (Estimated up to 4 Months)
Overall Survival (OS) | Baseline to Death from Any Cause (Estimated up to 6 Months)
Pharmacokinetics (PK): Systemic Clearance (CL) of LY287358 | Baseline to Study Completion (Estimated up to 4 Months)
Pharmacokinetics (PK): Volume of distribution (V) of LY287358 | Baseline to Study Completion (Estimated up to 4 Months)
PFS | Baseline to Measured Progressive Disease or Death from Any Cause (Estimated up to 6 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea